CLINICAL TRIAL: NCT03064425
Title: Understanding HIV Susceptibility in the Female Genital Tract
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 14-007
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Vaginal and blood sample collection — The researchers will obtain approximately 20 mL of blood from participants. Participants will also undergo a pelvic exam where a sample of cells will be collected from the cervix using two small cytobrushes. In addition, a cervicovaginal lavage will be collected using saline.

SUMMARY:
There is great variability in susceptibility from one person to another, and less than one in a hundred sexual exposures to HIV results in infection. In addition, some recent trial of methods to prevent HIV - including vaccines and microbicides - have actually increased HIV acquisition among trial participants for reasons that we do not fully understand. While we know that immune differences in the genital lining are an important determinant of whether a person is infected after a sexual HIV exposure, we don't know enough about these differences to be able to accurately assess a person's individual HIV risk. Therefore, the development of safe and non-invasive laboratory tests to estimate a person's susceptibility in the genital tract would be useful in clinical studies of new HIV prevention tools.

DETAILED DESCRIPTION:
Heterosexual intercourse is the most common mode of transmission of HIV, but the risk of HIV acquisition after exposure is so low that studies to assess HIV risk must have a huge sample size. The goal of this study is to assess the suitability of a prototype pseudovirus assay to identify early HIV target cells in the female genital tract, using cervical cytobrush samples collected from healthy women, and to optimize assay sensitivity.

This novel HIV entry assay may overcome the need for a large sample size by directly measuring how susceptible a person is by using a sample similar to a PAP test. The assay is performed on immune cells obtained from a cervical cytobrush and enables assessment of HIV cell entry within 24 hours. If the assay works, this technique may have the potential to assess the impact of clinical parameters such as stage of menstrual cycle, or sexually transmitted infections and their treatment on HIV susceptibility in the female genital tract. Therefore, the assay may serve as an important monitoring tool in clinical trials of HIV prevention, serving as an invaluable intermediate endpoint to assess HIV acquisition risk, rather than relying on actual participant HIV seroconversion/infection.

ELIGIBILITY:
Inclusion Criteria:

* women over the age of 18 years

Exclusion Criteria:

1. pregnant
2. actively menstruating
3. known HIV infection
4. genital ulceration or discharge on history or physical examination

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Non-pregnant women
Study Population: This study is recruiting healthy non-pregnant women from the St. Michael's Gynecology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
CD4 cell infection | Assay to be conducted within 24 hours of sample collection
  The absolute number of CD4+ cells per cytobrush that are infected by HIV

SECONDARY OUTCOMES:
Type of infected CD4 cells | Assay to be conducted within 24 hours of sample collection
  Nature of the CD4+ cells that are infected, ie: identification of immune characteristics that are associated with preferential HIV cell entry. Parameters to be assessed include immune activation markers and the expression of HIV coreceptors and integrins.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yudin, MD, Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: No